CLINICAL TRIAL: NCT03875963
Title: Performance of Antibiotic Impregnated Calcium Sulfate: A Prospective Randomized Controlled Trial
Brief Title: Antibiotic Loaded Calcium Sulfate RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided not to pursue the study.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Biocomposites Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5148
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Fracture Non Union; Infection
Keywords: Infection; Antibiotic bone cement; Tibia nonunion
MeSH Terms: conditions — Fractures, Ununited; Infections

STUDY DESIGN:
Intervention Model Description: The proposed study is a multi-centered, prospective, randomized controlled trial, comparing current standard of care for defect management to placement of antibiotic loaded Stimulan as a bone void filler in patients undergoing treatment of infected tibial defects or infected tibial nonunions.
Who Masked: Outcomes Assessor
Masking Description: Determination of union assessed by two independent assessors blinded to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic loaded bone filler (Experimental): Patients will undergo irrigation and debridement, surgical stabilization as required, and defect management by placement of antibiotic loaded Stimulan as a bone void filler [calcium sulfate bone void filler (10 cc of STIMULAN(R) Rapid Cure, Biocomposites Ltd, UK) combined with the following antibiotic combination: 1g Vancomycin, 240mg Tobramycin]. The concurrent use of antibiotics is at the discretion of the treating physician.
  Interventions: Other: Antibiotic loaded bone filler
- Standard of care (No Intervention): Current standard of care treatment for infected tibial defects or infected tibial nonunions includes treatment with irrigation and debridement, surgical stabilization as required, and defect management as required including placement of a polymethyl methacrylate spacer with or without antibiotics. A second procedure may or may not occur 6-8 weeks later with removal of the cement spacer and bone grafting into the preserved defect. Concurrent use of antibiotics is at the discretion of the treating physician.

INTERVENTIONS:
Other: Antibiotic loaded bone filler — Defect management by placement of antibiotic loaded Stimulan as a bone void filler [calcium sulfate bone void filler (10 cc of STIMULAN(R) Rapid Cure, Biocomposites Ltd, UK) combined with the following antibiotic combination: 1g Vancomycin, 240mg Tobramycin].
  Arms: Antibiotic loaded bone filler

SUMMARY:
This is a multi-centered, prospective, randomized controlled trial comparing current standard of care for defect management to placement of antibiotic loaded Stimulan as a bone void filler in patients undergoing treatment of infected tibial defects or infected tibial nonunions.

DETAILED DESCRIPTION:
There is a tremendous burden of disease associated with infected bone defects and infected nonunions and their management is challenging. Infected bone defects and nonunions have a profound clinical and economic impact and outcomes are limited by high rates of re-operation and poor functional outcomes. Reconstruction of infected bone defects or nonunions is difficult with multiple treatment options that may be considered. A comprehensive approach includes the treatment of infection, the management of dead space, skeletal stabilization, stimulation of soft tissue healing and healing of the bone defect or nonunion.

There is little evidence and a distinct lack of consensus regarding the definitive management of infected bone defects and infected nonunions. A two stage approach is still the gold standard for management and it remains unclear when alternative approaches should be considered. The first stage of the procedure includes adequate debridement, skeletal stabilization as required and placement of a polymethyl methacrylate cement spacer with or without antibiotics at the site of the bone defect. The second stage typically occurs between 6-8 weeks later with removal of the cement spacer and bone grafting into the preserved defect. There is no clear preferred management strategy and there remains a significant evidence gap.

There has been a significant interest in the use of bone graft substitutes for defect management as part of the management of infected bone defects and infected nonunions. The use of calcium sulfate as an alternative synthetic bone graft material has long been established (1-4), and the combination of calcium sulfate with antibiotics has been reported in the literature almost as long as antibiotics have been available (5, 6).

The clinical performance of calcium sulfate in combination with a single antibiotic, Tobramycin, is well documented (7, 8). However, in recent years, the use of calcium sulfate in combination with multiple antibiotics has grown in use as a means of providing protection from bacterial colonization by a wider variety of gram negative and gram positive pathogens (9-12). This study will evaluate the clinical performance of a high purity calcium sulfate bone void filler, STIMULAN® Rapid Cure. STIMULAN® Rapid Cure is intended to be gently packed into bony voids or gaps of the skeletal system (i.e., extremities, pelvis, and posterolateral spine). STIMULAN® Rapid Cure provides a bone graft substitute that resorbs and is replaced with bone during the healing process. STIMULAN® Rapid Cure is biodegradable and biocompatible and may be used at an infected site.

The proposed study is a multi-centered, prospective, randomized controlled trial, comparing current standard of care for defect management to placement of antibiotic loaded Stimulan as a bone void filler in patients undergoing treatment of infected tibial defects or infected tibial nonunions. Patients with an infected tibial bone defect or infected tibial nonunion meeting inclusion criteria will be randomized to receive either standard of care for defect management (Group A) or placement of antibiotic loaded Stimulan (10cc Stimulan Rapid Cure, 1g Vancomycin, 240mg Tobramycin) as a bone void filler (Group B), with a standardized intervention and post-intervention protocol.

ELIGIBILITY:
Inclusion Criteria:

* ≥16 years old.
* Isolated infected tibia defect or infected tibial nonunion (characterized by clinical symptoms present for greater than 90 days, the presence of necrotic bone, and bacteria cultured from prior procedures, surgical biopsy, or draining sinuses).

Exclusion Criteria:

* Presence of previous vascular injury or pathologic fracture
* Associated lower limb injuries that would interfere with rehabilitation or outcome
* Refusal to participate
* Inability to provide informed consent
* Inability to speak/understand or read English without a registered interpreter.
* Allergy or sensitivity to Vancomycin or Tobramycin

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Number of re-operations | 2 years post-injury
  Number of re-operations to obtain union or manage malunion, implant failure, or to eradicate infection.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  Pain measured using valid and reliable numeric pain rating scale. The scale measures the intensity of pain on a scale of 0 (meaning no pain) to 10 (worst pain). The scale asks the participant to rate the intensity of their pain in three ways -- their current pain level, their best pain level in the past 24 hours, and their worst pain level in the past 24 hours. The mean of all three scores is calculated by the research staff for a final average score. A lower score would indicate a better outcome, while a higher score would indicate a worse outcome.
Functional Index In Trauma (FIX-IT) Measure | Baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  The scale consists of two subscales - a weightbearing subscale and a pain subscale. The weight-baring subscale consists of two weight-bearing measures (Single Leg Score and Ambulation Score) and the pain subscale consists of two pain assessment measures (Palpation Score and Stress Score). Each of the four measures are rated on a scale from 0 to 3, with higher values representing a better outcome. For the weight bearing subscale, the Single Leg-Stand and the Ambulation Scores are added together, and for the pain subscale, the Palpation and the Stress Scores are added together for a total maximum score out of 6. The two subscales are added together at the end for a total maximum score of 12.
Patient reported outcomes | Baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  Short Musculoskeletal Function Assessment
EuroQol Group Quality of Life Scale with 5 Dimensions and 5 Levels (EQ-5D-5L) | Baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  The EuroQol5D-5L measures overall health and quality of life in 5 dimensions - Mobility, Self-care, Usual Activities, Pain/Discomfort, Anxiety/Depression. Each subscale is given a score from 0 to 4, with higher scores representing a worse outcome. The 5 subscale scores are added together for a total maximum score out of 20. There is one additional question which asks the participant to rate their overall perceived health today on a scale from 0 to 100 with 0 representing the worst health they can imagine and 100 representing the best health they can imagine.
Number of patients with complications | Baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  Complications assessed will include nonunion, malunion, leg length discrepancy, infection, wound healing problems, and drainage
Economic analysis | Baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  Ambulatory and Health Care Record to record economic burden on patient
Radiographic assessment | Baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months
  a) Anteroposterior and lateral tibial x-rays of all patients will be obtained at the standard follow-up intervals and will be blinded and scored by two established orthopaedic surgeons who are familiar with the RUST and modified RUST assessment scales b) Defect size pre-treatment will be measured using anteroposterior and lateral tibial x-rays

CONTACTS AND LOCATIONS:
Overall Officials: Emil Schemitsch, MD FRCS(C), Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] PELTIER LF. The use of plaster of paris to fill large defects in bone. Am J Surg. 1959 Mar;97(3):311-5. doi: 10.1016/0002-9610(59)90305-8. No abstract available. PMID 13627355
- [Background] PELTIER LF. The use of plaster of Paris to fill defects in bone. Clin Orthop. 1961;21:1-31. No abstract available. PMID 14485018
- [Background] PELTIER LF, BICKEL EY, LILLO R, THEIN MS. The use of plaster of paris to fill defects in bone. Ann Surg. 1957 Jul;146(1):61-9. doi: 10.1097/00000658-195707000-00007. No abstract available. PMID 13435702
- [Background] Peltier LF, Jones RH. Treatment of unicameral bone cysts by curettage and packing with plaster-of-Paris pellets. J Bone Joint Surg Am. 1978 Sep;60(6):820-2. PMID 701318
- [Background] KOVACEVIC B. [Problem of hematogenous osteomyelitis]. Langenbecks Arch Klin Chir Ver Dtsch Z Chir. 1953;276:432-43. No abstract available. Undetermined Language. PMID 13143827
- [Background] Fischer G, Seidler W. [Results in the treatment of osteomyelitic bone cavities using antibiotic gypsum medullary plombage]. Dtsch Gesundheitsw. 1971 Nov 4;26(45):2105-7. No abstract available. German. PMID 5145654
- [Background] McKee MD, Li-Bland EA, Wild LM, Schemitsch EH. A prospective, randomized clinical trial comparing an antibiotic-impregnated bioabsorbable bone substitute with standard antibiotic-impregnated cement beads in the treatment of chronic osteomyelitis and infected nonunion. J Orthop Trauma. 2010 Aug;24(8):483-90. doi: 10.1097/BOT.0b013e3181df91d9. PMID 20657257
- [Background] McKee MD, Wild LM, Schemitsch EH, Waddell JP. The use of an antibiotic-impregnated, osteoconductive, bioabsorbable bone substitute in the treatment of infected long bone defects: early results of a prospective trial. J Orthop Trauma. 2002 Oct;16(9):622-7. doi: 10.1097/00005131-200210000-00002. PMID 12368641
- [Background] Gauland C. Managing lower-extremity osteomyelitis locally with surgical debridement and synthetic calcium sulfate antibiotic tablets. Adv Skin Wound Care. 2011 Nov;24(11):515-23. doi: 10.1097/01.ASW.0000407647.12832.6c. PMID 22015750
- [Background] Jogia RM, Modha DE, Nisal K, Berrington R, Kong MF. Use of highly purified synthetic calcium sulfate impregnated with antibiotics for the management of diabetic foot ulcers complicated by osteomyelitis. Diabetes Care. 2015 May;38(5):e79-80. doi: 10.2337/dc14-3100. No abstract available. PMID 25908163